CLINICAL TRIAL: NCT07262333
Title: Safety and Pharmacokinetics of Single-dose Hydroxynidone Capsules in Patients With Renal Insufficiency
Brief Title: A Trial of Hydroxynidone Capsules in Single-dose Administration for Patients With Renal Insufficiency
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KDN-F351-202503
Record Dates: First submitted 2025-11-17; First posted 2025-12-03 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Renal Insufficiency Chronic
Keywords: Hydroxynidone
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — hydronidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (healthy individuals) (Experimental): On the morning of Day 1, take 90mg of hydronidone capsules on an empty stomach.
  Interventions: Drug: Hydronidone capsules
- The group of patients with mild renal insufficiency(eGFR 60~89 mL/min) (Experimental): On the morning of Day 1, take 90mg of hydronidone capsules on an empty stomach.
  Interventions: Drug: Hydronidone capsules
- The group of patients with moderate renal insufficiency(eGFR 30~59 mL/min) (Experimental): On the morning of Day 1, take 90mg of hydronidone capsules on an empty stomach.
  Interventions: Drug: Hydronidone capsules
- The group of patients with severe renal insufficiency(eGFR 15~29 mL/min) (Experimental): On the morning of Day 1, take 90mg of hydronidone capsules on an empty stomach.
  Interventions: Drug: Hydronidone capsules

INTERVENTIONS:
Drug: Hydronidone capsules — Take 90mg orally on an empty stomach on Day 1.

SUMMARY:
Hydronidone capsules are pyridinone-based small molecule compounds. Hydronidone has not been approved for commercial sale both domestically and internationally. The applicant has completed the preliminary Phase I and Phase II clinical trials. The results showed that Hydronidone is a safe and effective drug for treating liver fibrosis in chronic hepatitis B, and it has good safety and tolerability.

Based on the preliminary clinical research, a special population study has been initiated. The aim is to investigate the pharmacokinetic differences and safety of honginone capsules in patients with renal insufficiency and healthy subjects, in order to provide a basis for the clinical medication of patients with renal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* The subjects must meet all of the following criteria to be eligible for inclusion:
* (1) Healthy Chinese subjects, with an estimated glomerular filtration rate (absolute eGFR) meeting the following conditions: ≥ 90 mL/min and < 130 mL/min; (limited to healthy subjects)
* (2) Patients diagnosed with renal dysfunction, with the estimated glomerular filtration rate (absolute eGFR) for mild, moderate, and severe renal dysfunction meeting the following standards respectively: 1. Mild renal dysfunction 60-89 mL/min; 2. Moderate renal dysfunction 30-59 mL/min; 3. Severe renal dysfunction 15-29 mL/min; (limited to patients with renal dysfunction)
* (3) Age 18-70 years old, inclusive of 18 years and 70 years old;
* (4) Weight: Male ≥ 50 kg, female ≥ 45 kg, 18 ≤ BMI ≤ 28 (BMI = weight (kg) / height2 (m2));
* (5) During the 24 hours before the start of the trial to the end of the trial, the subjects agree to quit smoking, alcohol, fruit juices, caffeine, and tea;
* (6) Before the trial, they have fully understood the nature, significance, possible benefits, possible inconveniences, and potential risks of the trial, and voluntarily participated in this clinical trial, can communicate well with the researchers, comply with all the requirements of the entire study, and have the ability to understand and sign the written informed consent form.

Exclusion Criteria:

* The following conditions must be met for a subject to be eligible for this trial:
* (1) If the subject has participated in any other clinical trial within the three months prior to the trial;
* (2) If the subject has any disease that may affect the safety of the trial or the body's process of the drug, excluding renal insufficiency, including but not limited to: previous or existing diseases of the heart, liver, digestive tract, immune system and respiratory system (especially any gastrointestinal diseases that affect drug absorption, such as irritable bowel syndrome symptoms, intestinal diseases or inflammatory bowel disease history, active pathological bleeding (such as peptic ulcers), urticaria, epilepsy, allergic rhinitis, eczematous dermatitis, asthma, etc.); (limited to patients with renal insufficiency);
* (3) If the subject has any disease that may affect the safety of the trial or the body's process of the drug, including but not limited to: previous or existing diseases of the heart, liver, kidney, endocrine, digestive tract, immune system and respiratory system (especially cardiovascular diseases including those with cardiovascular disease risk, any gastrointestinal diseases that affect drug absorption (such as irritable bowel syndrome symptoms, intestinal diseases or inflammatory bowel disease history), active pathological bleeding (such as peptic ulcers), urticaria, epilepsy, allergic rhinitis, eczematous dermatitis, asthma, etc.); (limited to healthy subjects);
* (4) If the subject has an allergic constitution: if there is a history of allergy to two or more drugs (including the trial drug), food, or lactose intolerance;
* (5) If the subject has used any drugs that inhibit or induce the liver's metabolism of the drug within 28 days before taking the study drug (common liver enzyme inducers: barbiturates, carbamazepine, amiloride, griseofulvin, amitriptyline, phenytoin, grumet, rifampicin, dexamethasone; common liver enzyme inhibitors: chlorpromazine, cimetidine, ciprofloxacin, metronidazole, chloramphenicol, isoniazid, sulfonamide drugs);
* (6) If the subject has used drugs that inhibit or induce SULT and UGT enzymes within 7 days before taking the study drug and cannot stop the use;
* (7) If the subject cannot tolerate venipuncture and/or has a history of fainting or needle shock;
* (8) If the subject has long-term excessive consumption of tea, coffee or caffeinated beverages (more than 8 cups per day, 1 cup = 250 mL) in the past; or if within 24 hours before the first administration of the study drug, the subject consumed any food or beverage that inhibits or induces liver metabolic enzymes (such as grapefruit, mango, dragon fruit, grape juice, orange juice, etc., which contain rich flavonoids or citrus glycosides compounds); or if within 24 hours before the first administration of the study drug, the subject took any product containing alcohol;
* (9) If the subject has consumed blood or had a large amount of bleeding (more than 450 mL) within 3 months before the first administration of the study drug, or plans to donate blood or blood components during or after the study;
* (10) If the subject has donated blood or had a large amount of bleeding (more than 450 mL) within 3 months before the first administration of the study drug, or plans to donate blood or blood components during or after the study;
* (11) If the subject has acute diseases during the screening stage of the study or before taking the study drug;
* (12) If the subject has consumed foods or beverages that inhibit or induce liver metabolic enzymes within 24 hours before the first administration of the study drug (such as grapefruit, mango, dragon fruit, grape juice, orange juice, etc., which contain rich flavonoids or citrus glycosides compounds);
* (13) If the subject is pregnant or breastfeeding, and the subject (or their partner) has a pregnancy plan during and after the study, and does not agree to use non-drug measures for contraception during the study period;
* (14) (Medical Inquiry) Those who underwent surgery within three months prior to the screening period, or those planning to undergo surgery during the study period, and those who have undergone surgeries that may affect drug absorption, distribution, metabolism, and excretion;
* (15) Those with a history of drug use or drug abuse;
* (16) Those who smoked more than 5 cigarettes per day within 14 days prior to the screening, or those who cannot stop using any tobacco products during the trial;
* (17) Those who smoked or used any tobacco products during the screening to admission period;
* (18) Those whose physical examination, vital sign measurement, electrocardiogram examination, laboratory tests (urine and blood routine, coagulation function, blood pregnancy [only for women of childbearing age]) as determined by the researchers show abnormal results with clinical significance (excluding abnormalities caused by renal insufficiency). Abnormal liver function tests (ALT, AST, ALP, γ-GT, TP, Alb, A/G, T-BIL, D-BIL) indicate liver disease or liver damage; renal function tests with SCr > 400 µmol/L; abnormal blood electrolyte tests (K+, Na+, Cl-, Ca2+), indicating high potassium or a tendency towards acidosis; (for patients with renal insufficiency)
* (19) Those whose physical examination, vital sign measurement, electrocardiogram examination, laboratory tests [blood routine, urine routine, blood biochemistry, coagulation function, blood pregnancy (only for women of childbearing age)] as determined by the researchers show abnormal results with clinical significance; (for healthy subjects)
* (20) Those with positive nicotine test results;
* (21) Those with alcohol breath test results greater than 0.0 mg/100 ml;
* (22) Those with positive urine drug screening results;
* (23) Those with positive hepatitis B surface antigen, or hepatitis C antibody, or syphilis spirochete antibody, or HIV antibody test results positive;
* (24) Those who, as determined by the researchers, have any situation that may affect the subject's provision of informed consent or compliance with the trial protocol, or who participating in the trial may affect the trial results or their own safety.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-12-25 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
The plasma drug concentrations of hydronidone and its metabolites M3 and M4(AUC0-∞) | 48 hours after administration
The free plasma concentration of hydronidone | 48 hours after administration
The urine drug concentrations of hydronidone and its metabolites M3 and M4 | 48 hours after administration
The plasma drug concentrations of hydronidone and its metabolites M3 and M4(AUC%Extrap) | 48 hours after administration
The plasma drug concentrations of hydronidone and its metabolites M3 and M4( AUC0-t) | 48 hours after administration
The plasma drug concentrations of hydronidone and its metabolites M3 and M4(CL/F) | 48 hours after administration
The plasma drug concentrations of hydronidone and its metabolites M3 and M4(Vd/F) | 48 hours after administration
The plasma drug concentrations of hydronidone and its metabolites M3 and M4(Cmax) | 48 hours after administration
The plasma drug concentrations of hydronidone and its metabolites M3 and M4(T1/2) | 48 hours after administration
The plasma drug concentrations of hydronidone and its metabolites M3 and M4(λz) | 48 hours after administration
The plasma drug concentrations of hydronidone and its metabolites M3 and M4(Tmax) | 48 hours after administration

SECONDARY OUTCOMES:
Safety indicator: Any adverse event | 72 hours after administration
  Adverse Event (AE) is defined as any untoward medical occurrence during drug clinical trials, drug therapy, or medical procedures, regardless of its causal relationship to the drug used.
Safety indicator: B-ultrasound examination(liver) | 72 hours after administration
Safety indicator: B-ultrasound examination(gallbladder) | 72 hours after administration
Safety indicator: B-ultrasound examination(pancreas) | 72 hours after administration
Safety indicator: B-ultrasound examination(spleen) | 72 hours after administration
Safety indicator: B-ultrasound examination(kidneys) | 72 hours after administration
Safety indicators:12-lead electrocardiogram examination. | 72 hours after administration
  The 12-lead electrocardiogram records the electrical activity of the heart through 12 different lead positions, and is the most commonly used and fundamental non-invasive examination method for diagnosing heart diseases.A 12-lead ECG examines P waves, PR intervals, QRS complexes, ST segments, T waves, QT intervals, and other ECG waves and intervals.

CONTACTS AND LOCATIONS:
Overall Officials: shaojun Shi, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Hubei, Wuhan, China